CLINICAL TRIAL: NCT05092087
Title: Effects of Nutritional Counseling Regularity on the Risk of Cardiovascular Diseases
Status: Completed | Type: Observational
Sponsor: Taipei Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: N202103134
Record Dates: First submitted 2021-09-01; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-04

CONDITIONS: Cerebrovascular Disease
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group/ non-regularity group: those who completed 8 consultations by average interval time more than 3 weeks were in the non-regularity group
  Interventions: Behavioral: nutrition counseling
- test group/ regularity group: those who completed the consultations and interval time within in 3 weeks were in the higher regularity
  Interventions: Behavioral: nutrition counseling

INTERVENTIONS:
Behavioral: nutrition counseling — nutrition counseling

SUMMARY:
This study aims to investigate the frequency of personalized nutrition counseling's effect on individual cardiovascular risk factors. The study collected 110 to 150 cases data, including a regular blood test, blood glucose, blood lipid, liver panel, and inflammatory factors. The enrolled cases were classified into two groups according to the subjects' duration of consultation: those who completed the consultation and subsequent tests in >24 weeks were in the control group, whereas those who completed the consultation and subsequent tests in <24 weeks were in the test group. The effectiveness of nutrition consultation toward managing cardiovascular disease risk factors and its correlation with the subjects' frequency of following the consultations was analyzed using the pre- and post-consultation data. It was found that personalized nutrition consultation significantly improved the subjects' risk factors of cardiovascular diseases, and that the treatment group showed a greater improvement than the control group which who require over 24 weeks to complete all consultation sessions.

DETAILED DESCRIPTION:
The most of interventional studies on nutrition consultation have generally emphasized on the extent to which the diet composition can prevent chronic diseases or provide improvement. Although dietitians play an important role in health education for the primary prevention of chronic disease, their individuals dietary consultation results are mostly focused on weight loss and blood glucose control. However, the effectiveness of nutrition consultation on the prevention of chronic diseases, such as hyperlipidemia, hypertension and cardiovascular diseases, has few been studied. The effectiveness of dietary instructions provided to individuals by dietitians in primary health care institutes is yet to be validated with significant evidence. In addition, nutrition consultation methods, processes, and influencing factors on its results are seldom discussed. Therefore, this study aims to investigate the frequency of personalized nutrition counseling's effect on individual cardiovascular risk factors. The study collected1 10 to 150 cases data who aimed to prevent or improve chronic diseases and had completed eight times individualized nutrition consultations from Bon Vivant Health Lifestyle Management Center, and the pre- and post-consultation data, including a regular blood test, blood glucose, blood lipid, liver panel, and inflammatory factors, will be analyzed. Blood were drawn before and after the first and the last time consultation for biochemical tests; blood pressure and body composition was also measured for comparison. The enrolled cases will be classified into two groups according to the subjects' duration of consultation: those who completed the consultation and subsequent tests in >24 weeks were in the control group, whereas those who completed the consultation and subsequent tests in <24 weeks were in the test group. The effectiveness of nutrition consultation toward managing cardiovascular disease risk factors and its correlation with the subjects' frequency of following the consultations was analyzed using the pre- and post-consultation data. It was found that personalized nutrition consultation significantly improved the subjects' risk factors of cardiovascular diseases, and that the treatment group showed a greater improvement than the control group which who require over 24 weeks to complete all consultation sessions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 20
* Anyone of follow： body mass index > 24 systolic blood pressure > 120 mmHg diastolic blood pressure > 80 mmHg triglyceride > 150 mg/dL fasting blood glucose >100 mg/dL

Exclusion Criteria:

* Age <20
* pregnant
* Mental problem
* unable to do the measurement of body composition
* incomplete the nutritional counseling program

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who volunteer to pay and completed nutrition consultations from Bon-Vivant Health Lifestyle Management Center.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
body weight | baseline, pre-intervention
  body weight in kilograms
body weight | immediately after the intervention
  body weight in kilograms
height | baseline, pre-intervention
  height in meters
height | immediately after the intervention
  height in meters
body mass index | baseline, pre-intervention
  body mass index in kg/m^2
body mass index | immediately after the intervention
  body mass index in kg/m^2
body fat | baseline, pre-intervention
  body fat in ratio
body fat | immediately after the intervention
  body fat in ratio
The concentration of blood triglyceride | baseline, pre-intervention
  blood triglyceride in mg/dL
The concentration of blood total cholesterol | within one week after the intervention
  blood total cholesterol in mg/dL
The concentration of blood low density lipoprotein-cholesterol | baseline, pre-intervention
  blood blood low density lipoprotein-cholesterol in mg/dL
The concentration of blood low density lipoprotein-cholesterol | within one week after the intervention
  blood blood low density lipoprotein-cholesterol in mg/dL
The concentration of blood high density lipoprotein-cholesterol-cholesterol | baseline, pre-intervention
  blood high density lipoprotein-cholesterol in mg/dL
The concentration of blood high density lipoprotein-cholesterol-cholesterol | within one week after the intervention
  blood high density lipoprotein-cholesterol in mg/dL
The concentration of blood high sensitive C-reactive protein | baseline, pre-intervention
  blood high sensitive sensitive C-reactive protein in mg/L
The concentration of blood high sensitive C-reactive protein | within one week after the intervention
  blood high sensitive sensitive C-reactive protein in mg/L
The concentration of blood fasting glucose | baseline, pre-intervention
  blood fasting glucose in mg/dL
The concentration of blood fasting glucose | within one week after the intervention
  blood fasting glucose in mg/dL
blood HbA1C | baseline, pre-intervention
  blood HbA1C in percentage
blood HbA1C | within one week after the intervention
  blood HbA1C in percentage
The concentration of blood insulin | baseline, pre-intervention
  blood insulin in mg/dL
The concentration of blood insulin | within one week after the intervention
  blood insulin in mg/dL
The activity of blood aspartate aminotransferase | baseline, pre-intervention
  blood aspartate aminotransferase in U/L
The activity of blood aspartate aminotransferase | within one week after the intervention
  blood aspartate aminotransferase in U/L
The activity of blood alanine aminotransferase | baseline, pre-intervention
  blood alanine aminotransferase in U/L
The activity of blood alanine aminotransferase | within one week after the intervention
  blood alanine aminotransferase in U/L
The concentration of blood urinary nitrogen (BUN) | baseline, pre-intervention
  BUN in mg/L
The concentration of blood urinary nitrogen (BUN) | within one week after the intervention
  BUN in mg/L
The concentration of blood creatinine | baseline, pre-intervention
  BUN in mg/dL
The concentration of blood creatinine | within one week after the intervention
  BUN in mg/dL
The concentration of blood uric acid | baseline, pre-intervention
  blood uric acid in mg/dL
The concentration of blood uric acid | within one week after the intervention
  blood uric acid in mg/dL
The concentration of blood total protein | baseline, pre-intervention
  blood uric acid in mg/dL
The concentration of blood total protein | within one week after the intervention
  blood uric acid in mg/dL
The concentration of blood albumin | baseline, pre-intervention
  blood uric acid in mg/dL
The concentration of blood albumin | within one week after the intervention
  blood uric acid in mg/dL
The concentration of blood globulin | baseline, pre-intervention
  blood uric acid in mg/dL
The concentration of blood globulin | within one week after the intervention
  blood uric acid in mg/dL

CONTACTS AND LOCATIONS:
Overall Officials: Suh-Ching Yang, Study Chair — Taipei Medical University
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided